CLINICAL TRIAL: NCT05688150
Title: Prevalence and Associated Factors of Sarcopenia Among Elderly Patients in Osteoporosis Clinic
Status: Completed | Type: Observational
Sponsor: Kowloon Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Leung Hin Cheung, Principal Investigator, Kowloon Hospital, Hong Kong
Other Study IDs: KHRehab_LeungHC_1
Record Dates: First submitted 2022-12-21; First posted 2023-01-18 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Sarcopenia; Osteoporosis
Keywords: osteosarcopenia; sarcopenia; osteoporosis; geriatric medicine
MeSH Terms: conditions — Sarcopenia; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This was a cross-sectional study. Patients who attended the osteoporosis clinic of Kowloon Hospital from June to December 2022 were recruited.

Grip strength and appendicular skeletal muscle mass index were measured with a Jamar dynamometer and a bioimpedance analyser. Since most patients in our clinic are of Chinese ethnicity, the diagnostic criteria in the Consensus Update on Sarcopenia Diagnosis and Treatment by the Asian Working Group for Sarcopenia in 2019 was utilised. The diagnosis of sarcopenia was established by the presence of both low grip strength (Male: < 28 kg, Female < 18 kg) and low appendicular skeletal mass (Male: < 7.0 kg/m2, Female: < 5.7 kg/m2)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years old or above
* Diagnosed with osteoporosis by: Fragility fracture or T-score ≤-2.5 SDs at any site on DXA scan and;
* Able to read and write Chinese

Exclusion Criteria:

* Unable to maintain standing posture for bioimpedance analysis
* Modified Functional Ambulation Classification (MFAC) ≤ IV
* Incompetent in giving consent
* Unable to follow instructions
* Implanted with metal in any of four limbs
* Implanted with pacemaker, implantable cardioverter defibrillator or any other types of electrical device

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who attended the osteoporosis clinic of Kowloon Hospital from June to December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of Sarcopenia | June - December 2022
  The diagnosis of sarcopenia would be established by the co-existence of low grip strength and low appendicular skeletal muscle mass.
Grip strength | June - December 2022
  Grip strength would be measured with Jamar digital dynamometer.
Appendicular Skeletal Muscle Mass Index | June - December 2022
  Appendicular Skeletal Muscle Mass Index would be measured with bioimpedance analyzer.

SECONDARY OUTCOMES:
Association between BMI and Sarcopenia. | June - December 2022
  BMI would be measured on clinic attendance.
Association between Frailty and Sarcopenia. | June - December 2022
  Clinical Frailty Scale would be documented in clinical consultation.
Association between Charlson Comorbidities Index and Sarcopenia | June - December 2022
  Components of Charlson Comorbidities Index would be extracted from medical record.
Association between Bone Mineral Densities and Sarcopenia | June - December 2022
  Bone mineral densities of spine and neck of femur would be extracted from the report of dual-energy X-ray absorptiometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Kowloon Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882